CLINICAL TRIAL: NCT01724112
Title: 8-Week, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center Study of the Efficacy and Safety of LY2940094 Administered Once Daily in Patients With Major Depressive Disorder (MDD)
Brief Title: Study of the Efficacy and Safety of LY2940094 in Participants With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BlackThorn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14791; I5J-MC-NOAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-10-31; First posted 2012-11-09 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — LY2940094

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2940094 (Experimental): 40 mg administered orally as 1 capsule QD for 8 weeks.
  Interventions: Drug: LY2940094
- Placebo (Placebo Comparator): Administered orally as 1 capsule QD for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2940094 — Administered orally
  Arms: LY2940094
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This study will determine the efficacy, safety, and tolerability of a 40 milligrams (mg) once-daily (QD) dose of LY2940094 for 8 weeks in participants with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of MDD without psychotic features as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)
* Have clinically significant depressive symptoms defined by a GRID Hamilton Depression Rating Scale 17 (HAMD17) Total Score ≥20 at screening
* Body mass index (BMI) between 18 and 35 kilogram per square meter (kg/m²)

Exclusion Criteria:

* Have a current or previous diagnosis of bipolar I or II disorder, MDD with psychotic features, schizoaffective disorder, schizophrenia, or other psychotic disorder
* Currently meeting the criteria of treatment-resistant depression defined as ≥2 documented, failed treatment trials of adequate dose and duration with a registered antidepressant during the current depressive episode
* Had electroconvulsive treatment, transcranial magnetic stimulation, vagal nerve stimulation for symptoms of depression in the 6 months prior to screening
* Have any clinically significant medical or uncontrolled condition or circumstance prior to randomization that could affect participant safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 8 on the GRID Hamilton Depression Rating Scale 17 Item Version (GRID-HAMD17) Total Score | Baseline, Week 8

SECONDARY OUTCOMES:
Proportion of Participants Responding to Treatment | Baseline through Week 8
Proportion of Participants who Achieved Remission | Week 8
Change from Baseline to Week 8 in Maier-Philipp Subscale (MPS) Score | Baseline,Week 8
Clinical Global Impression - Improvement (CGI-I) Score at Week 8 | Week 8
Change from Baseline to Week 8 in the Clinical Global Impression - Severity (CGI-S) Score | Baseline, Week 8
Change from Baseline to Week 4 in the Hamilton Anxiety Rating Scale (HAM-A) Total Score | Baseline, Week 4
Change from Baseline to Week 8 in the Hospital Anxiety and Depression Scale (HADS) Score | Baseline, Week 8
Population Pharmacokinetic (PK) Model: Estimate of LY2940094 Area Under the Curve (AUC) | Baseline through 8 Weeks of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakland Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., University Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clinton, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington